CLINICAL TRIAL: NCT04614493
Title: Multisite Open-label Randomized Phase II Clinical Trial in Newly Diagnosed Glioblastoma Treated by Concurrent Temoradiation and Adjuvant Temozolomide +/- Ultrasound-induced Blood Brain Barrier Opening.
Brief Title: Innovative SonoCloud-9 Device for Blood Brain Barrier Opening in First Line Temozolomide Glioblastoma Patients.
Acronym: SonoFIRST
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200080; 2020-001488-10 (EudraCT Number)
Record Dates: First submitted 2020-10-21; First posted 2020-11-04 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Initial Radiological Diagnosis Eligible for Tumor Resection; Initial Radiological Diagnosis Compatible With Newly Diagnosed Glioblastoma (IDH Wild-type); Eligible for the Standard of Care Including Concurrent Temoradiation and Adjuvant Temozolomide
Keywords: Primary brain cancer; Glioblastoma; first line; Stupp protocol; Ultrasounds; Medical device; SC9
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound experimental arm (Experimental): Standard of Care + 15 Ultrasound BBB opening
  Interventions: Device: SonoCloud-9 (SC9) device; Drug: Temozolomide according Stupp protocol
- Control arm (Other): Standard of Care
  Interventions: Drug: Temozolomide according Stupp protocol

INTERVENTIONS:
Device: SonoCloud-9 (SC9) device — daily temozolomide (TMZ) during Radiation, followed by 6 months of adjuvant TMZ (5 days/months) with 6 concomitant Blood Brain Barrier opening sessions by ultrasound
  + 9 Blood Brain Barrier opening sessions by ultrasound without any associated drug
  Arms: Ultrasound experimental arm
Drug: Temozolomide according Stupp protocol — daily temozolomide (TMZ) during Radiation, followed by 6 months of adjuvant TMZ (5 days/months)

SUMMARY:
Glioblastoma (GBM) is an aggressive cancer with a progression-free survival (PFS) of 7 months and an overall survival (OS) of 15 months. Many therapeutic approaches have failed to improve the prognosis of patients to date. One of the main reasons is the presence of blood brain barrier (BBB) which limits therapeutic agents uptake in the brain. GBM is also considered to have a "cold" (unresponsive) immunological microenvironment due to factors released by the tumor and the presence of BBB limiting the transit of immune cells from the systemic circulation. Therefore, by-passing the BBB appears as a promising strategy.

The objective of the Phase II clinical trial, SonoFIRST, is to evaluate if the use of therapeutic ultrasound device, sonoCloud-9 (SC9) could improve the progression free survival of newly diagnosed GBM patients, treated by concurrent temoradiation and adjuvant temozolomide. The transient opening of the BBB by ultrasound with the SonoCloud-9 (SC9) device, predicts the increase in the penetration of temozolomide (TMZ) into the brain and the stimulation of cerebral immunity with the prospect of improving the survival of 160,000 new brain tumor patients each year in Europe and the United States.

DETAILED DESCRIPTION:
This will be an open-label, Phase 2, multicenter, double arm, randomized, interventional trial that will evaluate primarily the clinical efficacy of the device and will be to compare Progression Free Survival (PFS) between the standard of care treatment with concomitant ultrasound BBB opening versus standard of care alone. Glioblastoma (GBM) is the most common and aggressive primary brain cancer. Currently, prognosis is very poor, with a survival of about 15 months with current therapies. Although intensive treatments combining surgery, radiotherapy and chemotherapy, the prognosis of GBM patients remains poor. New treatment strategies are urgently needed.

In the brain, the presence of the blood-brain barrier (BBB) limits the uptake of therapeutic agents. To encounter this BBB issue, Professor Alexandre Carpentier and his team developed an ultrasound medical device (SonoCloud), implanted in the skull during surgery. This highly innovative technique temporarily permeates the BBB, increasing drug delivery to the brain by five times. The SonoCloud, a low-intensity pulsed ultrasound device developed by CarThera, is one of the major innovations in this field, as shown by the encouraging results obtained in studies in recurrent GBM.

The expected benefits of using the SonoCloud-9 experimental device prior to TMZ chemotherapy are the stabilization or reduction of GBM tumor volume on the one hand, and stabilization or improvement of the patient's neurological status on the other hand.

Participation in the clinical trial will contribute to a better understanding of the safety and efficacy of opening the BBB. It will be possible to determine whether the BBB opening using low-intensity pulsed ultrasound can be effective in treating GBM, in addition to the standard of care protocol.

ELIGIBILITY:
Inclusion Criteria :

1. Age ≥ 18 years , able and willing to give signed and informed consent. Inclusion for patients aged >70 years should be validated in neuro-oncology tumor board (RCP)
2. MRI with suspicion of GBM or Patient with a newly histologically proven IDHwt GBM by previous stereotaxic biopsy or king size opened biopsy
3. Karnofsky Performance Status ≥ 70
4. Patient eligible for a total or sub-total surgical tumor resection
5. Maximal tumor enhancement diameter at inclusion (pre surgery) ≤ 70 mm in T1W MRI
6. Patient eligible after surgery for the first line standard of care temoradiation and adjuvant TMZ (Stupp protocol, 54)
7. Patient with adequate organ and bone marrow function within 14 days prior to registration, as defined below:

   * Hemoglobin ≥ 10.0 g/dL
   * Leukocytes ≥ 3,000/L
   * Absolute neutrophil count ≥ 1,500/L
   * Platelets ≥ 100,000/L
   * Total bilirubin < 1.5 x ULN
   * AST(SGOT)/ALT(SPGT) ≤ 3 x institutional ULN
   * Alkaline phosphatase (ALP) < 3 x ULN
   * Normal creatine clearance ≥ 60 mL/minute.
   * Prothrombin time and partial thromboplastin time within institutional limits.
8. For women of childbearing potential, a negative pregnancy test before inclusion and a medically acceptable method of birth control used throughout the study are required. A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions applies: Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 1 month after the end of study visit
9. A male patient must agree to use contraception as detailed in this Protocol during the treatment period and for at least 6 months after the last cycle of TMZ; he must refrain from donating sperm during this period
10. Patient capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the Informed Consent Form (ICF) and in this protocol
11. Patient must be a beneficiary of or affiliated with a social security scheme

Exclusion Criteria :

1. Patients with multifocal tumor (unless all localized in a 70 mm diameter area accessible to ultrasound field) or located in posterior fossa tumor
2. Patient with diffuse FLAIR abnormalities attributable to Gliomatosis
3. Patients with evidence of uncontrolled intracranial pressure
4. Patients with uncontrolled epilepsy
5. Patients with medical need to continue antiplatelet or antithrombotic treatment
6. Pregnant or breastfeeding women (blood pregnancy test)
7. Patients with contra-indications to MRI or known sensitivity/allergy to gadolinium, or other intravascular contrast agents
8. Known history of hypersensitivity reactions to perflutren lipid microsphere components or to any of the inactive ingredients in Luminity®/Definity®
9. Patients with known intracranial aneurism, with and/or unremovable coils, clips, shunts, intravascular stents, wafer, non resorbable dura substitute, or reservoirs
10. Patients with an uncontrolled intercurrent illness or any pre-existing comorbidities that in the Investigator's opinion may prevent the implantation of the device or may impair the ability of the patient to receive treatment with SonoCloud or may be cofounding for evaluation of the clinical trial.
11. Patients with the following are not eligible:

    * Known arterial hypertension grade 3 or higher without adequate control on medications
    * Known or suspected unstable active or chronic infections requiring systemic treatment
    * Known significant cardiac disease: right-to-left shunts, Unstable angina pectoris, Symptomatic congestive heart failure, Unstable cardiac arrhythmia
    * Known significant pulmonary disease: severe pulmonary hypertension (pulmonary artery pressure > 90 mmHg), uncontrolled systemic hypertension, adult respiratory distress syndrome, or Pneumonitis
    * Known Severe renal failure
    * Known serious myelosuppression
    * Known Psychiatric illness/social situations that would limit compliance with study requirements
    * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
    * Known immunodeficiency disease or treatments (HIV)
    * Known viral or bacterial chronic/acute disease (potential blood borne infections that could result in meningitis or brain abscess)
12. Patients under judicial protection
13. Patients with any following prohibited treatments:

    * Any investigational medicinal product within 30 days prior to inclusion and during the study
    * Antibiotics with known neurotoxicity (eg, aminoglycosides, cephalosporin, quinolones), unless substitution is not possible,
    * Non-absorbable material (dura matter substitute, hemostatic agent…)
    * Any other drug according investigator to cause cerebral toxicity due to BBB opening
    * Contra-indications to temozolomide
    * Dacarbazine hypersensitivity
14. Implantation of the SC-9 not possible according to neurosurgeon (any patient morphological characteristics (e.g. skin thin thickness >9mm), which, from neurosurgeons' opinion, prevent implantation of the device or may impair the ability of the patient to receive treatment with SonoCloud, would be excluded)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-09-11 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS), PFS is defined as the time between randomization and disease progression which is the first documented tumor progression (per local Investigator assessment according to the RANO criteria) or death due to any cause. | Between randomisation and 18 months after the last inclusion.
  Progression will be assessed by local investigator according to the RANO criteria

SECONDARY OUTCOMES:
Overall Survival improvement (OS) | Between randomisation and 18 months after the last inclusion.
  OS is defined as the time from the date of randomization to the date of death due to any cause.
central review Progression Free Survival (crPFS) | Between randomisation and 18 months after the last inclusion.
  The central review Progression Free Survival is evaluated by a central assessment (independent imaging core lab) at the end of study and is defined as the time between randomization and tumor progression which is the first documented tumor progression according to the radiological RANO criteria or death due to any cause
immune Progression Free Survival (iPFS) | Between randomisation and 18 months after the last inclusion.
  The iPFS is evaluated according to iRANO (immune-related modifications / pseudo-progression ) criteria assessed by local investigator
Mean score of Patient quality of life preservation - EORTC Quality of Life Questionnaire C30 | Before surgery, pre-TemoRadiation visit, Cycle 1 (baseline after surgery/radiotherapy, 1 cycle = 28 days), Cycle 3, Cycle 6, Month 11 and Month 18, or until progression up to 18 months
  Quality of Life Questionnaire (QLQ) according to the European Organization for Research and Treatment of Cancer will be assessed by mean scores of the EORTC QLQ C-30 questionnaire (30 questions, score from 30 to 126) by local investigator or nurses and patient
Mean score Patient quality of life preservation - BN20 Quality of Life Questionnaire | Before surgery, pre-TemoRadiation visit, Cycle1 (baseline after surgery/radiotherapy, 1 cycle = 28 days), Cycle 3, Cycle 6, Month 11, Month 18, or until progression up to 18 months
  Quality of Life Questionnaire (QLQ) according to the European Organization for Research and Treatment of Cancer will be assessed will be assessed by means of the EORTC BN20 questionnaire (30 questions, score from 1 to 80) by local investigator or nurses and patient
Karnofsky Performance Status (KPS) | Before surgery, Surgery (+/- device implantation), pre-TemoRadiation visit, start and day 15 of each cycle (=28 days) from Cycle 1 to 6, Month 11, Month 13, Month 15, or until progression up to 18 months, new surgery (debulking or device explantation)
Mean score of Patient cognitive preservation | Before surgery, pre-TemoRadiation visit, Cycle1 (baseline after surgery/radiotherapy, 1 cycle = 28 days), Cycle 3, Cycle 6, Month 11, Month 18, or until progression up to 18 months
  Mini Mental Status Examination (30-point questionnaire, score from 1 to 30) mean score assessed by local investigator or nurses and patient
Visual analogic scale (VAS) Pain score from surgical area | Before surgery, pre-TemoRadiation visit, Cycle1 (baseline after surgery/radiotherapy, 1 cycle = 28 days), Cycle 3, Cycle 6, Month 11, Month 18, or until progression up to 18 months
  pain score from surgical area using visual analogic scale (score 0 to 10. Zero indicates the absence of pain, while 10 represents the most intense pain possible).
Esthetical | Before surgery, pre-TemoRadiation visit, Cycle1 (baseline after surgery/radiotherapy, 1 cycle = 28 days), Cycle 3, Cycle 6, Month 11, Month 18, or until progression up to 18 months
  score in self-confidence concerning esthetical dimension of surgical scar using esthetical comfort question equivalent to q39 of QLQ-BR23 questionnaire: Does your skull scar induce any esthetic burden to you?
  1. Not at all
  2. A little
  3. Quite a bit
  4. Very much
Safety : Type, frequency and severity of adverse events and serious adverse events | From inclusion to end of treatment, up to 18 months
  Safety confirmation of efficient blood brain barrier opening procedure with the SonoCloud-9 system. Safety confirmation is assessed by the frequency and severity of Adverse Events (AE) (incidence of AE summarized by system organ class and/or preferred term and severity) based on the Common Terminology Criteria for Adverse Events, version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed IDBAIH, MD, PhD, Principal Investigator — APHP-Sorbonne, Pitie Salpetriere Hospital, Paris
Locations (7):
- Katholieke Universiteit Leuven, Leuven, Belgium
- France (5):
  - Centre hospitalier Universitaire d'Angers, Angers
  - Groupe Hospitalier Saint-André, Bordeaux
  - Hospices Civils de Lyon, Hôpital Pierre Wertheimer, Bron
  - AP-HM, La Timone, Hôpital Universitaire, Marseille
  - APHP-Sorbonne, Pitié Salpêtrière Hospital, Paris
- Centre hospitalier universitaire vaudois CHUV, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carpentier A, Canney M, Vignot A, Reina V, Beccaria K, Horodyckid C, Karachi C, Leclercq D, Lafon C, Chapelon JY, Capelle L, Cornu P, Sanson M, Hoang-Xuan K, Delattre JY, Idbaih A. Clinical trial of blood-brain barrier disruption by pulsed ultrasound. Sci Transl Med. 2016 Jun 15;8(343):343re2. doi: 10.1126/scitranslmed.aaf6086. PMID 27306666
- [Background] Idbaih A, Canney M, Belin L, Desseaux C, Vignot A, Bouchoux G, Asquier N, Law-Ye B, Leclercq D, Bissery A, De Rycke Y, Trosch C, Capelle L, Sanson M, Hoang-Xuan K, Dehais C, Houillier C, Laigle-Donadey F, Mathon B, Andre A, Lafon C, Chapelon JY, Delattre JY, Carpentier A. Safety and Feasibility of Repeated and Transient Blood-Brain Barrier Disruption by Pulsed Ultrasound in Patients with Recurrent Glioblastoma. Clin Cancer Res. 2019 Jul 1;25(13):3793-3801. doi: 10.1158/1078-0432.CCR-18-3643. Epub 2019 Mar 19. PMID 30890548